CLINICAL TRIAL: NCT03762785
Title: Pharmacokinetics and Dynamics of Nebulized Dexmedetomidine in Preschool Children Undergoing Abdominal Cancer Surgery
Brief Title: Pharmacokinetics and Dynamics of Nebulized Dexmedetomidine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, lecturer of anesthesia, ICU and pain manegement, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 435
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Abdominal Cancer
Keywords: pharmacokinitics; nebulized; dexmedetomidine; preschool children

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nebulized dexmedetomidine 2ug/kg (Active Comparator): inhalation of dexmedetomidine in the dose of 2ug/kg by nebulization
  Interventions: Drug: nebulized Dexmedetomidine
- nebulized dexmedetomidine 3ug/kg (Active Comparator): inhalation of dexmedetomidine in the dose of 3ug/kg by nebulization
  Interventions: Drug: nebulized Dexmedetomidine

INTERVENTIONS:
Drug: nebulized Dexmedetomidine — inhalation of dexmedetomidine by nebulizer. the study drug will be prepared in 3 ml of 0.9% saline and will be administered by standard hospital jet nebulizer via face-mask with continuous flow of 100%oxygen at 6 l/m for 10 to 15 min
  Other Names: pharmacokinitics of nebulized dexmedetomidine

SUMMARY:
the aim of this study is to study the pharmacokinetics and dynamics of nebulized dexmetedomidine in children undergoing major abdominal cancer surgery.

DETAILED DESCRIPTION:
Inhalation of nebulized drug is an alternative route of administration that is relatively easy to set up, does not require venpuncture, but is associated with high bioavailability of the administered drug. Information on the pharmacokinetics of dexmedetomidine in the pediatric population is very limited, especially in children. To the best of investigators knowledge, there are no published reports on the pharmacokinetics of nebulized dexmedetomidine in children.

ELIGIBILITY:
Inclusion Criteria:

* child aged 2-7 years
* ASA I or II
* scheduled for abdominal surgery
* with average weight, height, normal serum albumin

Exclusion Criteria:

* patients with allergy to the study drug
* patients with significant organ dysfunction
* patients with cardiac arrhythmia
* patients with congenital heart disease
* use of psychotropic medication and mental retardation.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
pharmacokinitics of dexmedetomidine | at the basline and after the end of nebuization of the drug at 5 minutes,15 minutes,30 minutes, 45 minutes, 60 minutes, 90 minutes and 120 minutes
  serum level of dexmedetomidine

SECONDARY OUTCOMES:
sedation score | baseline and after end of the drug adminstration by 30 mininute
  Ramsy sedation score
  1 = Anxious or restless or both Unacceptable; increase sedation 2=Cooperative, orientated and tranquil Acceptable; no action necessary 3=Responding to commands Acceptable; no action necessary 4=Brisk response to stimulus Acceptable; no action necessary 5=Sluggish response to stimulus Unacceptable; monitor respiratory status and sedation level until stable at 2 or 3 6= No response to stimulus Unacceptable; monitor respiratory status and sedation level until stable at 2 or 3

CONTACTS AND LOCATIONS:
Overall Officials: Shereen M Kamal, Lecturer, Principal Investigator — Ministry of higher education
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt